CLINICAL TRIAL: NCT04210687
Title: A Randomized Comparison Between Trapeziectomy and Trapeziometacarpal Limited Excision for Thumb Base Osteoarthritis
Brief Title: Trapeziectomy vs. Trapeziometacarpal Limited Excision for Thumb Base Osteoarthritis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Maria Wilcke, Prinicipal investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TEvsTLE
Record Dates: First submitted 2019-12-19; First posted 2019-12-26 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Thumb Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Trapeziectomy (Active Comparator): Standard simple trapeziectomy, no pins.
  Interventions: Procedure: Trapeziectomy
- trapeziometacarpal limited excision (Active Comparator): Trapeziometacarpal limited excision; Narrow pseudarthrosis of the trapeziometacarpal joint.
  Interventions: Procedure: trapeziometacarpal limited excision

INTERVENTIONS:
Procedure: trapeziometacarpal limited excision — Narrow pseudarthrosis CMC1
  Arms: trapeziometacarpal limited excision
Procedure: Trapeziectomy — Simple trapeziectomy
  Arms: Trapeziectomy

SUMMARY:
A randomized comparison between trapeziectomy and trapeziometacarpal limited excision for thumb base osteoarthritis in 90 patients.

ELIGIBILITY:
Inclusion Criteria:

* Painful osteoarthritis in the thumb base and radiological arthritis (Eaton Littler class 2-3) and clinical signs of thumb base osteoarthritis (pain at palpation of the thumb base joint and pain during grinding test).
* Pain at rest.
* Conservative treatment >6 months (activity modification, splinting, painkillers or thumb base steroid or PRP injection)

Exclusion Criteria:

* Rheumatoid arthritis.
* Ongoing infection in the hand or wrist. -
* History of gout or pseudo gout.
* Inability to co-operate with the follow-up protocol (language difficulties, severe psychiatric disorder, cognitive impairment, drug addiction).
* Intra-articular injection in the affected joint within 6 months.
* Eaton Littler class 4 (STT joint involved).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-03-09 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in pain on load NRS (numerical rating scale) | Preoperatively, 1, 3 and 5 years postoperatively
  Change in rated pain on load from preoperatively to 1, 3 and 5 years postoperatively

SECONDARY OUTCOMES:
Change in Nelson Thumb score | Preoperatively, 1, 3 and 5 years postoperatively
  0-100 p, higher score = less disability
Change in EQ-5D | 1, 3 and 5 years postoperatively
  Weight mean value: 0=dead, 1= healthy
Change in DASH - Disability of the Arm, Shoulder and Hand | Preoperatively, 1, 3 and 5 years postoperatively
  0-100 p, higher score = more disability
Change in PRWHE - Patient-Rated Wrist and Hand Evaluation | Preoperatively, 1, 3 and 5 years postoperatively
  0-100 p, higher score = more disability
Change in HADS - Change hospital Anxiety and Depression score | Preoperatively, 1, 3 and 5 years postoperatively
  2 subscores for anxiety (0-21P) and depression (0-21p), higher score = worse
Change in PCS - Pain Catastrophizing Score | Preoperatively, 1, 3 and 5 years postoperatively
  0-52, higher score = more pain catastrophizing
Change in Thumb base motion | Preoperatively, 1, 3 and 5 years postoperatively
  radial and palmar abduction of the first metacarpal (degrees).
Change in thumb strength | Preoperatively, 1, 3 and 5 years postoperatively
  Key pinch and pinch strength (Kg)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Wilcke, MD PhD, Principal Investigator — Karolinska Instituet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No